CLINICAL TRIAL: NCT00433082
Title: Effect of Fasting With Two Meals on Inflammatory Markers of Metabolic Syndrome
Brief Title: Metabolic Syndrome and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Free Islamic University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1345104
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome,Ramadan,Fasting,Inflammatory markers,; Iran
MeSH Terms: conditions — Metabolic Syndrome

INTERVENTIONS:
Behavioral: Ramadan Fasting

SUMMARY:
The metabolic syndrome has been recognized as a proinflammatory state. It has been shown that many different diets such as Mediterranean diet, DASH diet, Foods with low glycemic index and low saturated fat diet, independent of weight loss, may be effective in improving the metabolic syndrome. Our objective was to evaluate the effect of Ramadan fasting on High-sensitive C-reactive protein (hs-CRP) and fibrinogen levels in metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Males with metabolic syndrome

Exclusion Criteria:

* Conditions with insulin resistance including;
* Type 2 diabetes mellitus,
* Infections,
* Stresses,
* Uremia,
* Acromegaly,
* Glucocorticoid excess,
* Hypertension ,
* Cirrhosis and
* Any addiction or drug therapy and conditions witch cause changes in hs-CRP and fibrinogen levels including infection, trauma, infarction, inflammatory arthritis, various neoplasm and liver diseases.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-08; Study Completion 2006-11

PRIMARY OUTCOMES:
Measuring inflammatory markers in metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi, MD, Principal Investigator — Islamic Free University of Medical Science